CLINICAL TRIAL: NCT05726084
Title: Multicentre, Double-blind, Randomized, Prospective, Placebo-controlled Trial to Assess the Immunogenicity, Efficacy and Safety of the Coronavirus Vaccine in Healthy Volunteers Aged 18 Years and Older
Brief Title: Immunogenicity, Efficacy and Safety Trial of the Convacell Vaccine in Healthy Volunteers Aged 18 Years and Older
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Petersburg Research Institute of Vaccines and Sera (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 02-COVAC-02/22
Record Dates: First submitted 2023-01-17; First posted 2023-02-13 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: COVID-19; Coronavirus Infections; Respiratory Tract Infections; COVID-19 Respiratory Infection
Keywords: COVID-19; cellular immunity; nucleocapsid protein; recombinant vaccine; SPbSRIVS; SARS-CoV-2; Convacell
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Convacell, 1 dose (Stage IIb) (Experimental): Participants (230) will be vaccinated Convacell Vaccine, recombinant subunit vaccine for prevention of coronavirus infection, once intramuscularly. A cohort of participants will be allocated (115 participants) for evaluating cell-mediated immunity parameters.
  Interventions: Biological: Subunit recombinant vaccine for the prevention of coronavirus infection
- Convacell, 2 doses (Stage IIb) (Experimental): Participants (230) will be vaccinated Convacell Vaccine, recombinant subunit vaccine for prevention of coronavirus infection, twice intramuscularly. A cohort of participants will be allocated (115 participants) for evaluating cell-mediated immunity parameters.
  Interventions: Biological: Subunit recombinant vaccine for the prevention of coronavirus infection
- Convacell, chosen regimen (Stage III) (Experimental): Participants (10 562) will be vaccinated Convacell Vaccine, recombinant subunit vaccine for prevention of coronavirus infection, the regimen chosen in Stage IIb intramuscularly.
  Interventions: Biological: Subunit recombinant vaccine for the prevention of coronavirus infection
- Placebo, chosen regimen (Stage III) (Placebo Comparator): Participants (5 282) will be vaccinated Placebo, the regimen chosen in Stage IIb intramuscularly.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Subunit recombinant vaccine for the prevention of coronavirus infection — solution for intramuscular injection, 0.5 ml
  Other Names: Convacell
  Arms: Convacell, 1 dose (Stage IIb); Convacell, 2 doses (Stage IIb); Convacell, chosen regimen (Stage III)
Biological: Placebo — solution for intramuscular injection, 0.5 ml
  Arms: Placebo, chosen regimen (Stage III)

SUMMARY:
The goal of this clinical trial is to assess the immunogenicity, efficacy and safety of the Convacell vaccine in healthy adult volunteers aged 18 years and older. The main questions it aims to answer are:

* To assess the immunogenicity and safety of single and double dose intramuscular administration of the Convacell vaccine;
* To assess the epidemiological effectiveness of the Convacell vaccine in the prevention of SARS-CoV-2 infection and development of severe COVID-19 compared with placebo when single or double intramuscular injection.

DETAILED DESCRIPTION:
The trial will be conducted in two stages (Stage IIb and Stage III).

• Stage IIb

Participants will be vaccinated one dose or two doses of the Convacell vaccine. Investigators will compare one dose and two doses groups and will choose the best vaccine dosage regimen in terms of immunogenicity and safety.

• Stage III

Participants will be vaccinated the Convacell vaccine or Placebo. Investigators will use the dosage regimen chosen in IIb stage.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 Years and Older
* Written informed consent of the volunteer to participate in the clinical trial (in paper or electronic form)
* BMI within the range of 18.5 ≤ BWI ≤ 30 kg/m2 with the body weight of not less than 55 kg for men, not less than 45 kg for women and not more than 100 kg for volunteers of both sexes
* Absence of clinically significant (according to the investigator) deviations from the reference values of clinical, laboratory and instrumental methods of examination at screening
* Hemodynamic and other vital signs are within normal limits (reference intervals are 60-90 beats/min at rest for HR, up to 22 per minute for RR, body temperature from 35.5 to 36.9 °C; systolic blood pressure (SBP) is considered normal in the range of 100-139 mmHg, diastolic blood pressure (DBP) - in the range of 60-89 mmHg)
* Volunteers able to fulfill requirements of the Protocol (i.e., fill in the electronic patient's diary, come to follow-up visits)
* Abstinence from alcohol from the start of screening until completion of Visit 7 procedures (day 42 ± 2) - for stage 2b
* For fertile women - a negative result of the pregnancy test and consent to observe adequate methods of contraception during the trial and at least two months after vaccination
* For fertile men - consent to observe adequate methods of contraception during the trial and at least two months after vaccination, except for men after vasectomy with documented azoospermia, and their sexual partners should use methods of contraception that ensure more than 90% reliability or be incapable of conception after a surgical sterilization or have a natural menopause for at least 2 years
* Throughout the study, the opportunity to use own smartphone with the ability to fill in the electronic patient's diary

Exclusion Criteria:

* History of influenza or acute respiratory viral infection (ARVI) within 2 months before the start of the trial;
* A serious post-vaccination reaction (temperature above 40 °C, hyperemia or edema more than 8 cm in diameter) or complications (collapse or shock-like condition that developed within 48 hours after vaccination; convulsions accompanied or not accompanied by a fever due to any previous vaccination);
* Fever, cough, and shortness of breath within 30 days before vaccination;
* History of COVID-19 within 6 months before screening;
* The level of IgG antibodies to the SARS-CoV-2 N-protein according to semi-quantitative test (Architect, Abbott) ≥ 3 (positivity rate) at screening;
* Positive result of the COVID-19 PCR test or antigen COVID-19 test (rapid test);
* Body temperature ≥ 37,3°C.
* History of allergies;
* Any vaccination within 30 days before the screening;
* History of leukemia, tuberculosis, cancer, autoimmune diseases;
* History of Quincke's edema;
* Positive blood test results for HIV, syphilis, hepatitis B/C according to the examination during the screening period (only for Stage IIb) or according to the history (for Stage III). It is acceptable to use the results of previously performed tests, if their prescription does not exceed 60 days before the date of the screening or based on history;
* Volunteers who received immunoglobulin during the last three months before the trial;
* History of long-term use (more than 14 days) of immunosuppressants or other immunomodulatory drugs for six months before the trial;
* Treatment with glucocorticosteroids, including in small doses, as well as local use of drugs containing steroids (> 10 mg of prednisolone or its equivalent for more than 14 days before the screening);
* History of any confirmed or suspected immunosuppressive or immunodeficiency condition;
* History of splenectomy;
* History of chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems, the gastrointestinal tract, liver, kidneys, hematopoietic or immune systems, mental disease in the acute stage or in the decompensation stage (according to history and / or examination on the screening);
* Transfusion of blood or blood components within 4 months before screening;
* Any acute infectious diseases during the screening period or past illnesses within 3 months before the screening visit, any chronic infectious diseases in the acute stage during the screening period;
* Consumption of more than 10 units of alcohol per week or history of alcohol addiction, drug addiction or abuse of pharmaceutical products;
* Smoking of more than 10 cigarettes per day;
* Participation in another clinical trial within the last 90 days;
* Pregnancy or lactation;
* Coagulopathy, hemophilia, bleeding disorder;
* Participation in previous clinical trials of the Convacell vaccine, a subunit recombinant vaccine for the prevention of coronavirus infection caused by SARS-CoV-2 virus, or any other vaccines to prevent coronavirus infection caused by the virus SARS-CoV-2 for 6 months before screening;
* History of anticovid plasma use;
* Vaccination against COVID-19 within 6 months before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16304 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in titer of IgG antibodies to N-protein of SARS-CoV-2 (Stage IIb) | Days 0, 42
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
Frequency of symptomatic COVID-19 with laboratory-confirmed infection within 6 months after vaccination compared with the placebo group (Stage III) | Days 0-180 (6 months)
  Laboratory confirmation of SARS-CoV-2 infection in accordance with current clinical guidelines can be a PCR study or an antigen test of a swab from the nasopharynx or oropharynx.
  The symptomatic form of COVID-19 is the presence of at least one of the following symptoms: fever/chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body pain, headache, loss of the sense of taste or smell, sore throat, nasal congestion or runny nose, nausea or vomiting, diarrhea.
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.

SECONDARY OUTCOMES:
Change in titer of IgM antibodies to N-protein of SARS-CoV-2 on day 42 after initial vaccination (Stage IIb) | Days 0, 42
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
Proportion of SARS-CoV-2 seropositive participants on day 42 after initial vaccination (Stage IIb) | Days 0, 42
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
Change in titer of IgG antibodies to N-protein of SARS-CoV-2 on day 42 after initial vaccination (Stage IIb) | Days 0, 42
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
The frequency of seroconversion (appearance of specific antibodies to SARS-CoV-2 N-protein) on day 42 after initial vaccination (Stage IIb) | Days 0, 42
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
Change from Baseline in the Mean Specifically Sensitized T-lymphocytes (Stage IIb) | Days 0, 42
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
Number of volunteers hospitalized with COVID-19 (Stage IIb) | through trial Stage IIb; Days 0-49
  * Total number of SARS-CoV-2 infection cases (laboratory-confirmed)
  * Total number of COVID-19 cases (laboratory-confirmed)
  * Total number of COVID-19 related deaths
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
Frequency of laboratory confirmed asymptomatic SARS-CoV-2 infections within 6 months. after initial vaccination compared with the placebo group (Stage III) | Days 0-180 (6 months)
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
Frequency of laboratory-confirmed severe COVID-19 (Stage III) | Days 0-180 (6 months)
  Frequency of laboratory-confirmed severe COVID-19 in accordance with current criteria
  * RR > 30/min
  * Blood oxygen saturation (SpO2) ≤ 93%
  * Oxygenation index (PaO2 /FiO2) ≤ 300 mmHg
  * Decreased level of consciousness, agitation
  * Unstable hemodynamics (systolic arterial pressure [SBP] less than 90 mm Hg. or diastolic blood pressure [DBP] less than 60 mmHg, diuresis less than 20 ml/hour)
  * Lung changes on computed tomography (CT) or radiographs typical for a viral lesion
  * Arterial blood lactate > 2 mmol/l
  * Assessment on a quick scale (quick Sequential Organ Failure Assessment, qSOFA) > 2 points
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
Overall frequency of all AEs/SAEs (Stage IIb and III) | through trial Stage IIb (Days 0-49), through trial Stage III (Days 0-196)
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
Overall frequency of all AEs/SAEs associated with the study drug (Stage IIb and III) | through trial Stage IIb (Days 0-49), through trial Stage III (Days 0-196)
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
The frequency of local post-vaccination reactions at the injection site (Stage IIb and III) | Days 0-7 after initial vaccination and revaccination
  * Erythema at the injection site (presence/absence);
  * Soreness (presence/absence), including assessment duration of preservation of pain and its intensity: weak, moderate, strong;
  * Edema (presence/absence), including diameter infiltrate assessment: weak (up to 2.5 cm), medium (from 2.6 to 5 cm), strong (more than 5 cm or the presence of lymphangitis) reactions;
  * Enlargement of regional lymph nodes (presence/absence);
  * Induration at the injection site (presence/absence);
  * Itching at the injection site (presence/absence).
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
The frequency of systemic post-vaccination reactions at the injection site (Stage IIb and III) | Days 0-7 after initial vaccination and revaccination
  * Increase in body temperature, including an assessment fever severity: mild (37.3-37.5°C), moderate (37.6-38.5°С) and strong (> 38.5°С);
  * Chills;
  * Deterioration of general health, malaise;
  * Headache;
  * Dizziness;
  * Loss of appetite;
  * Insomnia;
  * Nausea, Vomiting, Dyspepsia;
  * Diarrhea;
  * Body pain or muscle weakness;
  * Sweating;
  * Pain in the joints;
  * Pain in the abdomen;
  * Convulsions;
  * Myalgia;
  * Enlargement of regional lymph nodes.
  * Changes in the side of the mucous membranes, the presence of papules, vesicles, erosions.
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
The frequency of local post-vaccination reactions at the injection site (Stage IIb and III) | Days 0-21 after initial vaccination and revaccination
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
Frequency of systemic post-vaccination reactions (Stage IIb and III) | Days 0-42 after initial vaccination
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
The frequency of toxic post-vaccination complications (Stage IIb and III) | through trial Stage IIb (Days 0-49), through trial Stage III (Days 0-196)
  Septic conditions, generalized infection.
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
The frequency of allergic post-vaccination complications (Stage IIb and III) | through trial Stage IIb (Days 0-49), through trial Stage III (Days 0-196)
  Polymorphous eruption, angioedema, arthralgia, anaphylactic shock.
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
The frequency of neurological post-vaccination complications (Stage IIb and III) | through trial Stage IIb (Days 0-49), through trial Stage III (Days 0-196)
  Encephalitis, neuritis, polyneuritis.
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
The presence of allergic reactions (Stage IIb and III) | through trial Stage IIb (Days 0-49), through trial Stage III (Days 0-196)
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
Сhange in white blood cell count and relative white blood cell count (Stage IIb) | Day 0 (screening), day 28 ± 2 (visit 4)
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
Сhange in neutrophils count and relative neutrophils count (Stage IIb) | Day 0 (screening), day 28 ± 2 (visit 4)
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
Сhange in lymphocytes count and relative lymphocytes count (Stage IIb) | Day 0 (screening), day 28 ± 2 (visit 4)
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
Сhange in monocyte count and relative monocyte count (Stage IIb) | Day 0 (screening), day 28 ± 2 (visit 4)
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
Сhange in the IgE level (Stage IIb) | Day 0 (screening), day 28 ± 2 (visit 4)
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.
The proportion of participants with delayed post-vaccination reactions (percent) (Stage IIb and III) | through trial Stage IIb (Days 0-49), through trial Stage III (Days 0-196)
  Outcome Measure is analyzed separately in the 18-60 and >60 age subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Ellina Ruzanova, Study Director — St. Petersburg Research Institute of Vaccines and Sera
Locations (6):
- Russia (6):
  - Limited Liability Company "OLLA-MED", Moscow
  - State budgetary health care institution of the city of Moscow "City Clinical Hospital No. 24 of the Department of Health of the City of Moscow", Moscow
  - Limited Liability Company "Scientific Research Center Eco-Safety", Saint Petersburg
  - St. Petersburg State Budgetary Health Institution "City Polyclinic No. 117", Saint Petersburg
  - Limited Liability Company "Otkrytaya Meditsina", Tolyatti
  - Limited Liability Company "Meditsinskiy Diagnosticheskiy Tsentr", Yaroslavl